CLINICAL TRIAL: NCT03431558
Title: Can Bovine Lactoferrin Prevent Neonatal Infections in Low Birth Weight Babies in Karachi, Sindh, Pakistan.
Brief Title: Bovine Lactoferrin and Neonatal Survival in Low Birth Weight Babies.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: University of Sydney (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr Shabina Ariff, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SLAB
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Neonatal Sepsis; Necrotizing Enterocolitis
Keywords: Bovine Lactoferrin, Neonatal infection, Low Birth Weight
MeSH Terms: conditions — Neonatal Sepsis; Enterocolitis, Necrotizing

STUDY DESIGN:
Intervention Model Description: Group 1: bLF (150 mg) will be administered after 48 hours of age with a single daily dose mixed with milk (preferentially breast milk otherwise premature formula milk).
  Group 2: bLF will be administered (300mg) after 48 hours of life with a single daily dose mixed with milk (preferentially breast milk otherwise premature formula milk).
  Group 3: Placebo will be administered after 48 hours of life (Placebo will be physically identical to the bLF mixed with breast milk or premature formula milk).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be carried out by Data management unit and all investigators /dispensers and participants will be masked to the randomization.
  Clinical Trial Unit (CTU) of the Aga khan university will dispense the randomized supplemnt/placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): bLF (Bovine Lactoferrin plus Glucan D 99.4%) Dose: 150 mg Frequency: a single daily dose mixed with milk (preferentially breast milk otherwise formula milk).
  Duration: 1 month
  Interventions: Combination Product: bLF (Bovine lactoferrin)
- Group 2 (Experimental): bLF (Bovine Lactoferrin plus Glucan D 99.4%) Dose: 300mg Frequency: a single daily dose mixed with milk (preferentially breast milk otherwise formula milk).
  Duration: 1 month
  Interventions: Combination Product: bLF (Bovine lactoferrin)
- Group 3 (Placebo Comparator): Placebo: Only Glucan-D (99.4% glucoseDose: 150 mg Frequency: a single daily dose mixed with milk (preferentially breast milk otherwise formula milk).
  Duration: 1 month
  Interventions: Drug: Glucon-D 99.4% (Placebo)

INTERVENTIONS:
Combination Product: bLF (Bovine lactoferrin) — BLF administration in two different strengths (150 & 300mg) will be given on the third day of life with a single daily dose mixed with milk for 1 month.
  Other Names: bLF
  Arms: Group 1; Group 2
Drug: Glucon-D 99.4% (Placebo) — This group will be given 100mg Glucon-D (99.4% glucose) placebo which will be similar in shape, color to the bLF.
  Other Names: Placebo
  Arms: Group 3

SUMMARY:
Pakistan has the third highest number of neonatal deaths worldwide. During the last two decades (1990-2013), neonatal mortality rate in the country has declined by only 1.0% per year. Severe infection is the second most leading cause of neonatal mortality, account for 28% of all deaths in Pakistan. Majority of neonatal deaths occur in infants who LBW (birth weight <2500g) and LBW comprises of both preterm / small for gestational age newborns. Breastfeeding helps protect infants from infections by serving as a source of nutrition uncontaminated by environmental pathogens. The protection is due to the multiple anti-infective, anti-inflammatory, and immuno regulatory factors transmitted through milk including secretory antibodies, glycan's, Lactoferrin, leukocytes, cytokines & other components produced by the mother's immune system.

Reduction in neonatal infections and deaths is the aim of this study. The study is being conducted at the Aga Khan University in collaboration with University of Sydney.

DETAILED DESCRIPTION:
Globally, severe infection is the second leading cause of neonatal mortality. It is one of the indirect leading causes of death in a world. According to Annual report, 28% neonatal deaths were due to preterm baby, 26% due to severe infection , 23% due to asphyxia and 7% neonatal tetanus. Every year, three - fourth deaths occurred in first week and four million babies die each year within first four weeks of birth, whereas, 99% of cases were reported by low and middle income countries.Severe infections are the second major cause of death among neonates in Pakistan. Breastfeeding helps to protect infants from infections due to the multiple anti-infective, anti-inflammatory, and immuno regulatory factors such as secretory antibodies, glycan, Lactoferrin etc. Lactoferrin, the second most abundant protein in human milk has multiple putative functions. A trial in Italy found that the incidence of late-onset sepsis and sepsis related deaths were significantly lower in very LBW infants who were given daily (Bovine Lactoferrin) bLF compared to placebo. One small trial from India, found there was a 79% reduction in neonatal infections in LBW infants who received daily bovine Lactoferrin (bLF) from birth until 28 days. Evidence gaps remain about the appropriate daily prophylactic dose, the optimal method to deliver, and the effectiveness of bLF to prevent neonatal sepsis in LBW infants in low & middle-income countries.The overall goal of the project is to improve newborn survival among low birth weight (LBW) Pakistani infants through provision of a daily prophylactic dose of bLF. The project aim is to prevent neonatal infections, as opposed to the current approach which treats neonatal infections when they occur. The current approach depends on early detection of infections in newborns through post-natal care and treatment with antibiotics, with the potential risk of inappropriate use of antibiotics.A two stage study will be conducted including formative research followed by RCT to evaluate the appropriate daily dose of bLF. At the end of the study the investigators will have developed and tested an appropriate method to deliver bLF to newborns at home & identified the most appropriate dose of bLF to prevent neonatal sepsis in LBW newborns.

This study will be conducted at the Aga Khan University and Hospital, Karachi in two phases. A qualitative study will be conducted followed by a RCT. 300 LBW new born babies will be recruited;all standard operating procedures will be followed for administration of bLF to the neonates. Each arm of the study will be allocated 100 newborns.

ELIGIBILITY:
Inclusion Criteria:

Neonates with:

birth weight ≤ 2500 g and ≥ 1000 grams. gestational age ≥ to 28 +0 weeks to 36+6. family planned on staying in the study area for at least 1 month • parents/ caretaker willing to provide consent. newborn initiated enteral feeding via (gavage feeding with expressed breast milk or formula, direct breast feeding or cup and spoon feeding at or within 48 hours of birth.)

Exclusion Criteria:

Neonate with congenital anomalies. early-onset sepsis. birth weight less than 1000 g. gestational age less than or equal to 27weeks+6 days. history of Chorioamnionitis or maternal group B streptococcus colonization. Reversed or absent end-diastolic flow on maternal umbilical artery Doppler where available.

Ages: 48 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Late onset sepsis (LOS) in Low Birth Weight. | 1 month
  Reduction in late onset sepsis (LOS) in Low Birth Weight babies.
Optimal dosage of bLF | 1 month
  Deduce optimal dosage of bLF in LBW babies.

SECONDARY OUTCOMES:
Necrotizing Enterocolitis in LBW babies | 1 month
  Incidence of Necrotizing Enterocolitis in Low Birth Weight babies
Neonatal Mortality at 1 month of life. | 1 month
  Incidence of Neonatal Mortality at 1 month of life.

CONTACTS AND LOCATIONS:
Overall Officials: Shabina Ariff, MBBS,FCPS, Principal Investigator — Aga Khan University; Michael J Dibley, MB BS, MPH, Study Chair — University of Sydney; Almas Aamir, MSC, Study Director — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan A, Kinney MV, Hazir T, Hafeez A, Wall SN, Ali N, Lawn JE, Badar A, Khan AA, Uzma Q, Bhutta ZA; Pakistan Newborn Change and Future Analysis Group. Newborn survival in Pakistan: a decade of change and future implications. Health Policy Plan. 2012 Jul;27 Suppl 3:iii72-87. doi: 10.1093/heapol/czs047. PMID 22692418
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Hug L, Sharrow D, You D. Levels & trends in child mortality: report 2017. Estimates developed by the UN Inter-agency Group for Child Mortality Estimation. 2017.
- [Background] Farnaud S, Evans RW. Lactoferrin--a multifunctional protein with antimicrobial properties. Mol Immunol. 2003 Nov;40(7):395-405. doi: 10.1016/s0161-5890(03)00152-4. PMID 14568385
- [Background] Anderson BF, Baker HM, Dodson EJ, Norris GE, Rumball SV, Waters JM, Baker EN. Structure of human lactoferrin at 3.2-A resolution. Proc Natl Acad Sci U S A. 1987 Apr;84(7):1769-73. doi: 10.1073/pnas.84.7.1769. PMID 3470756
- [Background] The World Bank. Mortality rate, neonatal (per 1,000 live births) [29/02/2016]. Available from: http://data.worldbank.org/indicator/SH.DYN.NMRT.
- [Background] Kramer MS. Determinants of low birth weight: methodological assessment and meta-analysis. Bull World Health Organ. 1987;65(5):663-737. PMID 3322602
- [Background] Rahman S, Hameed A, Roghani MT, Ullah Z. Multidrug resistant neonatal sepsis in Peshawar, Pakistan. Arch Dis Child Fetal Neonatal Ed. 2002 Jul;87(1):F52-4. doi: 10.1136/fn.87.1.f52. PMID 12091293
- [Background] Morrow AL, Rangel JM. Human milk protection against infectious diarrhea: implications for prevention and clinical care. Semin Pediatr Infect Dis. 2004 Oct;15(4):221-8. doi: 10.1053/j.spid.2004.07.002. PMID 15494945
- [Derived] Ariff S, Soofi S, Aamir A, D'Almeida M, Aziz Ali A, Alam A, Dibley M. Bovine Lactoferrin to Prevent Neonatal Infections in Low-Birth-Weight Newborns in Pakistan: Protocol for a Three-Arm Double-Blind Randomized Controlled Trial. JMIR Res Protoc. 2021 Mar 11;10(3):e23994. doi: 10.2196/23994. PMID 33704071
- See also: The World Bank Mortality rate ,Neonatal (per,1000 live births) 29/02/2016 — http://data.worldbank.org/indicator/SH.DYN.NMRT
- See also: United.Nations Sustainable development goals — http://www.un.org/sustainabledevelopment/health